CLINICAL TRIAL: NCT04655222
Title: Non-interventional Safety Study to Investigate Pregnancy Outcomes in Female Patients Exposed to SC Peginterferon Beta-1a and IM Interferon Beta-1a Reported in a German Patient Support Program
Brief Title: Study to Investigate Pregnancy Outcomes in Female Participants Exposed to Subcutaneous (SC) Peginterferon Beta-1a and Intramuscular (IM) Interferon Beta-1a Reported in a German Participant Support Program
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-PEG-11650
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- All Participants: Pregnant Multiple Sclerosis (MS) participants treated with SC interferon beta therapy or an IM interferon beta therapy in the German PSP of the MSSC.
  Interventions: Drug: Interferon Beta Therapy

INTERVENTIONS:
Drug: Interferon Beta Therapy — Administered as specified in the treatment arm.

SUMMARY:
The primary objective(s) of the study is to evaluate the impact of exposure to SC Peginterferon beta-1a or IM Interferon beta-1a before and during pregnancy on pregnancy outcome in female participants who had registered in the German Patient Support Program (PSP) and of whom a pregnancy report and pregnancy outcome report is available.

The secondary objectives of this study are applicable for a subpopulation of the above-mentioned population, i.e. for participants of whom data on a standardized questionnaire collected during a telephone interview is available.

DETAILED DESCRIPTION:
This is an observational study with focus on existing pregnancy reporting forms (retrospective part) and a patient's questionnaire which is completed at a single point of time (prospective part). Main data source for the retrospective data (from 2014 until December 2019) will be captured from multiple sclerosis service-center (MSSC) database, i.e. the entered pregnancy report (to be completed as soon as pregnancy becomes known) and pregnancy outcomes report (to be completed after completion of pregnancy).

Prospective data (December 2020 to 31 March 2021) will be captured as standardized ePDF questionnaire completed during telephone interview. If the pregnancy report or the pregnancy outcome report is incomplete, i.e. the data above was not collected, the open questions will be addressed during a telephone interview performed by the MSSC and the new information will be entered into the MSCC database. The patient questionnaire will be completed at a single point of time during the telephone interview performed by the MSSC.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed relapsing-remitting multiple sclerosis (RRMS) or clinically isolated syndrome (CIS) (CIS indication only applicable for interferon beta-1a)
* Exposure to either SC Peginterferon beta-1a therapy or an IM Interferon beta-1a therapy before or during pregnancy
* Registered in the PSP of the multiple sclerosis service- center (MSSC) and agreed in writing to the privacy policy of the registration form
* Reported pregnancy data (pregnancy report and pregnancy outcome report) available at MSSC. Note: only pregnancy data (i.e. obtained until 15 October 2020) will be considered.
* Pregnancy outcome in the retrospectively collected data was a live birth

Exclusion Criteria: Any criteria that does not fulfil the above-mentioned inclusion criteria.

NOTE: Other protocol defined Inclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All female participants treated with SC Peginterferon beta-1a therapy or IM Interferon beta-1a therapy who fulfil the inclusion criteria are eligible to participate in the study.
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Live Births Without Congenital Anomalies | up to end of study (4 months)
Percentage of Participants With Live Births With Congenital Anomalies | up to end of study (4 months)
Percentage of Participants With Ectopic Pregnancies | 8 weeks of gestation
Percentage of Participants With Spontaneous Abortions | up to 22 weeks of gestation
  A spontaneous abortion is defined as fetal death before 22 weeks of gestation.
Percentage of Participants With Elective Abortions | up to Week 20 of gestation
Percentage of Participants With Preterm Births | up to 37 weeks of gestation
  A preterm birth is a birth before 37 completed weeks of gestation.
Percentage of Participants With Stillbirths | from 22 week up to 39 weeks of gestation
  A still birth is defined as fetal death at >22 weeks gestation.

SECONDARY OUTCOMES:
Average Weight of the Children | From Birth up to Month 48
Average Length of the Children | From Birth up to Month 48
Average Head Circumference of the Children | From Birth up to Month 48
Percentage of Abnormalities Diagnosed During Pediatric Check-ups | up to Month 48
Percentage of Women Discontinued Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy During Pregnancy | up to 39 weeks of gestation
Time to Discontinuation of Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy in Relation to Beginning of Pregnancy | up to 39 weeks of gestation
Percentage of Women Starting Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy During Pregnancy | up to 39 weeks of gestation
Time to Start Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy in Relation to Beginning of Pregnancy | up to 39 weeks of gestation
Percentage of Women Restarting Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy After Birth | up to end of study (4 months)
Time to Restart Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy in Relation to Birth | up to end of study (4 months)
Percentage of Women Starting Another Multiple Sclerosis (MS) Therapy During/After Pregnancy | up to end of study (4 months)
Time to Start Another MS Therapy During/After Pregnancy in Relation to Birth | up to end of study (4 months)
Percentage of Women Using Other Therapies During Pregnancy | up to 39 weeks of gestation
Percentage of Multiple Sclerosis Relapses in Women with Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy Before, During and After Pregnancy | up to end of study (4 months)
Change From Baseline Expanded Disability Status Scale (EDSS) During and After Pregnancy to Expanded Disability Status Scale (EDSS) Before Pregnancy | Week 0 up to Week 39 of gestation
  EDSS is based on a standardized neurological exam and focuses on symptoms that commonly occur in multiple sclerosis (MS). Scores range from 0.0 (normal) to 10.0 (death due to MS).
Number of Women Breastfeeding Under Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy | up to end of study (4 months)
Duration of Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy Exposed Breastfeeding | up to end of study (4 months)
Time to First Multiple Sclerosis (MS) Relapse After Introduction of the First Supplemental Feedings in Women With Subcutaneous Peginterferon Beta-1a or Intramuscular Interferon Beta-1a Therapy During Lactation | up to end of study (4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Klehmet J, Begus-Nahrmann Y, Taipale K, Niemczyk G, Rehberg-Weber K. Pregnancy outcomes in female multiple sclerosis patients exposed to intramuscular interferon beta-1a or peginterferon beta-1a reported in a German Patient Support Programme - results from the non-interventional post-authorization safety study PRIMA. Ther Adv Neurol Disord. 2023 Dec 15;16:17562864231214041. doi: 10.1177/17562864231214041. eCollection 2023. PMID 38107443
- [Derived] Klehmet J, Begus-Nahrmann Y, Taipale K, Niemczyk G, Rehberg-Weber K. Impact of interferon beta exposure on birth outcome and child development - Results from the post-authorisation safety study PRIMA. Mult Scler Relat Disord. 2023 Sep;77:104844. doi: 10.1016/j.msard.2023.104844. Epub 2023 Jun 24. PMID 37393802